CLINICAL TRIAL: NCT01452399
Title: A Randomized Controlled Trial of Routine Shave Margins vs. Standard Partial Mastectomy in Breast Cancer Patients
Brief Title: A Randomized Controlled Trial of Routine Shave Margins Versus Standard Partial Mastectomy in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1107008825
Record Dates: First submitted 2011-09-29; First posted 2011-10-14 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shave Margins (Experimental)
  Interventions: Procedure: Shave margins
- No shave margins (Active Comparator)
  Interventions: Procedure: No Shave Margins

INTERVENTIONS:
Procedure: Shave margins — Partial mastectomy with shave margins.
  Arms: Shave Margins
Procedure: No Shave Margins — Partial mastectomy without shave margins.
  Arms: No shave margins

SUMMARY:
This research study is designed to look at whether the routine use of shave margins (by taking extra tissue at the time of partial mastectomy surgery) will reduce the chances of having positive surgical margins requiring another surgical procedure, and whether this affects the long-term chances of getting cancer back in your breast.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer, stage 0-3, deemed a surgically appropriate candidate for partial mastectomy with planned procedure for the same.
2. Women ≥ 18 years of age.
3. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have received previous neoadjuvant chemotherapy
2. Patients who require a total mastectomy
3. Known metastatic breast cancer.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Optimal surgical treatment | 12 months
  To determine whether routine shave margins in breast cancer patients undergoing partial mastectomy will result in more optimal surgical treatment of breast cancer patients, as defined by reduced positive margin rates

SECONDARY OUTCOMES:
Cosmesis | 12 months
  To determine the effect of routine shave margins on cosmesis
Operative time | 12 months
  To determine the effect of routine shave margins on the time in the operating suite.
Volume of tissue resected | 12 months
  To determine the effect of routine shave margins on the volume of tissue resected.

CONTACTS AND LOCATIONS:
Overall Officials: Anees Chagpar, M.D., Principal Investigator — The Breast Center -- Smilow Cancer Hospital at Yale-New Haven
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Chagpar AB, Horowitz NR, Killelea BK, Tsangaris T, Longley P, Grizzle S, Loftus M, Li F, Butler M, Stavris K, Yao X, Harigopal M, Bossuyt V, Lannin DR, Pusztai L, Davidoff AJ, Gross CP. Economic Impact of Routine Cavity Margins Versus Standard Partial Mastectomy in Breast Cancer Patients: Results of a Randomized Controlled Trial. Ann Surg. 2017 Jan;265(1):39-44. doi: 10.1097/SLA.0000000000001799. PMID 27192352
- [Derived] Chagpar AB, Killelea BK, Tsangaris TN, Butler M, Stavris K, Li F, Yao X, Bossuyt V, Harigopal M, Lannin DR, Pusztai L, Horowitz NR. A Randomized, Controlled Trial of Cavity Shave Margins in Breast Cancer. N Engl J Med. 2015 Aug 6;373(6):503-10. doi: 10.1056/NEJMoa1504473. Epub 2015 May 30. PMID 26028131